CLINICAL TRIAL: NCT03251690
Title: Switching Tenofovir/Emtricitabine/Efavirenz to Tenofovir/Emtricitabine/Rilpivirine Versus Continuing Tenofovir/Emtricitabine/Efavirenz in HIV1-infected Patients With Complete Virological Suppression
Brief Title: Switching TDF/FTC/EFV to TDF/FTC/RPV VS Continuing TDF/FTC/EFV in HIV Patients With Complete Virological Suppression
Acronym: STEREOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID09-59-06
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Anti-Retroviral Agents; Efavirenz; HIV-1-infection; Sustained Virologic Response; Dyslipidemias; Rilpivirine
MeSH Terms: conditions — Dyslipidemias | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Switching TDF/FTC/EFV to TDF/FTC/RPV (Experimental): Switching from Tenofovir 300 mg/day + Emtricitabine 200 mg/day + Efavirenz 600 mg/day (once daily) to Tenofovir 300 mg/day + Emtricitabine 200 mg/day + Rilpivirine 25 mg/day (once daily) Intervention: Tenofovir/Emtricitabine/Rilpivirine
  Interventions: Drug: Tenofovir/Emtricitabine/Rilpivirine
- Continuing TDF/FTC/EFV (Active Comparator): Continuing Tenofovir 300 mg/day + Emtricitabine 200 mg/day + Efavirenz 600 mg/day Intervention: Tenofovir/Emtricitabine/Efavirenz
  Interventions: Drug: Tenofovir/Emtricitabine/Efavirenz

INTERVENTIONS:
Drug: Tenofovir/Emtricitabine/Rilpivirine — Tenofovir/Emtricitabine/Rilpivirine to compare the non-inferiority of efficacy and adverse effects to Tenofovir/Emtricitabine/Efavirenz in patients with virological suppression
  Other Names: TDF/FTC/RPV
  Arms: Switching TDF/FTC/EFV to TDF/FTC/RPV
Drug: Tenofovir/Emtricitabine/Efavirenz — as a active comparator
  Other Names: TDF/FTC/EFV
  Arms: Continuing TDF/FTC/EFV

SUMMARY:
According to the Thai National Guidelines for Treatment of HIV/AIDS 2014, the recommended first line ART regimen was 2 NRTIs backbone, TDF and FTC; plus 1 NNRTI, EFV, with RPV as an alternative one. Most of the randomized-controlled studies, including ECHO and THRIVE, showed the non-inferiority of RPV compared with EFV in naive cases. But there were not much randomized-controlled trials for changing from other NRTI to RPV in patients who currently on another ART, especially in Thailand. Moreover, the concerned adverse effects of dyslipidemia and neurological symptoms were better in RPV-based than EFV-based regimen. Finally, the cost-effectiveness and universal coverage are also the benefit of RPV over EFV in term of economics.

DETAILED DESCRIPTION:
According to the Thai National Guidelines for Treatment of HIV/AIDS 2014, the recommended first line ART (Anti-retroviral therapy) regimen was 2 NRTIs (nucleoside reverse transcriptase inhibitors) backbone, which are TDF (Tenofovir) and FTC (Emtricitabine); plus 1 NNRTI (non-nucleoside reverse transcriptase inhibitor), which is EFV (Efavirenz), with RPV (Rilpivirine) as an alternative in this class of drug.

Most of the randomized-controlled studies, including ECHO (Rilpivirine versus efavirenz with tenofovir and emtricitabine in treatment-naive adults infected with HIV-1) and THRIVE (Rilpivirine versus efavirenz with two background nucleoside or nucleotide reverse transcriptase inhibitors in treatment-naive adults infected with HIV-1), the major trials about RPV, showed the non-inferiority in efficacy of RPV compared with that of EFV in treatment-naive cases with blood HIV viral load less than 500,000 copies/mL. But there were not many trials focusing on changing the ART-regimens from other NRTI to RPV in patients who currently on another ART, especially in randomized-controlled design. There were some studies comparing continuing current regimens versus changing to Rilpivirine-based regimens, but they didn't exclusively select the homogeneous drug components. In Thailand, study of changing to Rilpivirine-based regimens was primarily designed to evaluate the adverse outcome about dyslipidemia, whereas efficacy was a secondary outcome. Most studies, the concerned adverse effects of dyslipidemia and neurological symptoms were better in RPV-based than EFV-based regimen. Finally, the cost-effectiveness and universal coverage are also the benefit of RPV over EFV in term of economics.

Therefore, we design this study to evaluate the efficacy; in term of non-inferiority, of the newer, safer, and cheaper drug, Rilpivirine, to Efavirenz, the general-use drug with acceptable efficacy, in the virological-suppressed patients currently on ART. Besides, we also assess the adverse outcomes and factors associated with successful or failure of treatment. In addition, we can have more backup data in term of national economics.

ELIGIBILITY:
Inclusion Criteria:

* on TDF/FTC/EFV for more than 3 months
* Blood HIV RNA viral load <50 copies/mL
* CD4+ count >200 cells/mm3
* eligible to sign the informed consent

Exclusion Criteria:

* history of NRTI resistance
* on medication that potentially interact with study drug
* denied to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2016-10-27 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Sustained virological response | 12 months
  maintain the undetectable HIV viral load

SECONDARY OUTCOMES:
Lipid adverse outcome | 12 months
  Different in blood lipid profiles, including triglycerides, cholesterol, HDL, and LDL
Neurological adverse outcome | 12 months
  Neurological adverse events such as dizziness
Cost -saving after switching regimens | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Sirichai Wiriyatanakorn, MD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Ramathibodi Hospital, Mahidol University; Somneuk Sungkanuparp, MD, Principal Investigator — Department of Internal Medicine, Faculty of Medicine, Ramathibodi Hospital, Mahidol University

REFERENCES:
- [Background] Thai AIDS Society. Thailand National Guidelines on HIV/AIDS Treatment and Prevention 2014. Nontaburi: Bureau of AIDS, TB, and STIs, 2014.
- [Result] Molina JM, Cahn P, Grinsztejn B, Lazzarin A, Mills A, Saag M, Supparatpinyo K, Walmsley S, Crauwels H, Rimsky LT, Vanveggel S, Boven K; ECHO study group. Rilpivirine versus efavirenz with tenofovir and emtricitabine in treatment-naive adults infected with HIV-1 (ECHO): a phase 3 randomised double-blind active-controlled trial. Lancet. 2011 Jul 16;378(9787):238-46. doi: 10.1016/S0140-6736(11)60936-7. PMID 21763936
- [Result] Cohen CJ, Andrade-Villanueva J, Clotet B, Fourie J, Johnson MA, Ruxrungtham K, Wu H, Zorrilla C, Crauwels H, Rimsky LT, Vanveggel S, Boven K; THRIVE study group. Rilpivirine versus efavirenz with two background nucleoside or nucleotide reverse transcriptase inhibitors in treatment-naive adults infected with HIV-1 (THRIVE): a phase 3, randomised, non-inferiority trial. Lancet. 2011 Jul 16;378(9787):229-37. doi: 10.1016/S0140-6736(11)60983-5. PMID 21763935
- [Result] Thamrongwonglert P, Chetchotisakd P, Anunnatsiri S, Mootsikapun P. Improvement of lipid profiles when switching from efavirenz to rilpivirine in HIV-infected patients with dyslipidemia. HIV Clin Trials. 2016 Feb;17(1):12-6. doi: 10.1080/15284336.2015.1112480. Epub 2016 Jan 7. PMID 26739573
- [Result] Gianotti N, Poli A, Nozza S, Spagnuolo V, Tambussi G, Bossolasco S, Cinque P, Maillard M, Cernuschi M, Galli L, Lazzarin A, Castagna A. Efficacy and safety in clinical practice of a rilpivirine, tenofovir and emtricitabine single-tablet regimen in virologically suppressed HIV-positive patients on stable antiretroviral therapy. J Int AIDS Soc. 2015 Jul 30;18(1):20037. doi: 10.7448/IAS.18.1.20037. eCollection 2015. PMID 26232000